CLINICAL TRIAL: NCT06483919
Title: The Predictive Value of Proteome Profiling for Brain Metastasis in Limited-Stage Small-Cell Lung Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: Jinming Yu (Other)
Responsible Party: Sponsor-Investigator, Jinming Yu, Director of the hospital, Shandong Cancer Hospital and Institute
Organization: Shandong Cancer Hospital and Institute (Other)
Other Study IDs: LS-SCLC-BM
Record Dates: First submitted 2024-06-26; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Small-cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SCLC patients with brain metastasis
- SCLC patients without brain metastasis

SUMMARY:
This study aims to evaluate the predictive value of proteome profiling for brain metastasis in limited-stage small-cell lung cancer

DETAILED DESCRIPTION:
Small-cell lung cancer (SCLC) constitutes approximately 15% of all lung cancer cases and is characterized by a highly aggressive disease course and poor prognosis. The brain is the most common metastatic site of SCLC, and it is also an important cause of high mortality. More than 20% of SCLC patients have developed brain metastasis (BM) at the first diagnosis. Prophylactic cranial irradiation (PCI), as an essential part of the treatment of limited-stage small-cell lung cancer (LS-SCLC), inevitably leads to neurotoxicity. Therefore, there is an urgent need for a convenient and effective prediction model to realize the early prediction of SCLC brain metastasis. Patients at high risk of brain metastases were treated with individualized PCI.

In the current study, the investigators have analyzed the proteome profiling using Data-independent Acquisition mass spectrometry (DIA-MS) method in formalin-fixed paraffin-embedded (FFPE) tissues from patients with limited-stage small-cell lung cancer. The prognostic biomarkers were developed based on machine learning in the non-PCI group. Patients in the non-PCI group were classified into modeling cohort and external validation cohort . Furthermore, the prognostic value of the candidate biomarkers be evaluated in a prospective cohort . Based on the brain metastasis model, patients were divided into high- and low-risk groups. The benefit value of PCI was analyzed in high-risk and low-risk groups.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years old
2. Histological / pathologic proved limited-stage small-cell lung cancer
3. Achieved a complete response (CR) or partial response (PR) after first-line CRT

Exclusion Criteria:

1. Simultaneous participation in another clinical trial
2. Brain MRI was not performed during treatment and follow-up
3. The follow-up time was less than 2 years
4. Patients presenting with other known malignancies for which they are receiving treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Limited-stage small-cell lung cancer
Sampling Method: Non-Probability Sample
Enrollment: 228 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-01-30 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
Brain metastases free survival | 2 years
  The length of time after the ending of primary treatment that the patient survives without any brain metastases signs or symptoms

SECONDARY OUTCOMES:
Overall survival | 2 years
  The length of time after the ending of primary treatment that the patient survives.

CONTACTS AND LOCATIONS:
Overall Officials: Xiangjiao Meng, PhD, Study Director — Shandong Cancer Hospital and Institute
Locations (1):
- Shandong Cancer Hospital and Institute, Jinan, Shandong, China